CLINICAL TRIAL: NCT05686161
Title: A Randomized, Single-blind, Parallel Controlled Trial to Evaluate the Immunogenicity ,Safety,Efficacy of A Heterologous Booster Dose With SW-BIC-213, in Previously Vaccinated Subjects Against COVID-19 With Two Inactivated COVID-19 Vaccine Doses Compared to a Booster Dose With Pfizer of Sinopharmin Adults
Brief Title: mRNA Booster Vaccine(SW-BIC-213) Compared With Pfizer andSinopharm Against Emerging VOCs
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stemirna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SWC310-1
Record Dates: First submitted 2022-12-20; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2022-10

CONDITIONS: Immunogenicity; Safety; Efficacy
Keywords: new generation mRNA vaccine

STUDY DESIGN:
Intervention Model Description: a randomized observer-blinded parallel controlled trial#Experimental group#mRNA vaccine# and positive control group#inactive vaccine#
Who Masked: Participant, Investigator
Masking Description: This study uses an observer-blinded design, and the investigators and participants will all remain blinded before unblinding and do not know which group the participant belongs to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A single 25 μg dose mRNA vaccine SW-BIC-213 (Experimental): Intervention Name :COVID-19 mRNA vaccine Type :Investigational Vaccine Dose :Formulation mRNA Unit Dose Strength(s) :0.5ml; Dosage Level(s) :0.25ml; Route of Administration: injection Intramuscular
  Interventions: Biological: SW-BIC-213;SARS-Cov-2.
- A third dose of COVID-19 Inactivated vaccine (Active Comparator): Intervention Name: COVID-19 Inactivated Vaccine Type : Control Vaccine Dose :Inactive Unit Dose Strength(s) : 0.5ml; Route of Administration: injection Intramuscular
  Interventions: Biological: Sinopharm (BIBP);SARS-Cov-2.
- A single 30μg dose mRNA vaccine Pfizer(BNT162b2) (Active Comparator): Type :mRNA COVID -19 vaccine - Pfizer(BNT162b2) Dose :Formulation mRNA Unit Dose Strength(s) :30ug; Dosage Level(s) :0.3ml; Route of Administration: injection Intramuscular
  Interventions: Biological: Pfizer(BNT162b2);SARS-Cov-2.

INTERVENTIONS:
Biological: SW-BIC-213;SARS-Cov-2. — The study will be performed in people receiving two doses of Sinopharm vaccine over 180 days (± 30 days) after the second dose prior to enrollment. The three study groups who will receive the booster dose will be assigned as follows:
  Subjects (N≈600) Group 1: (N≈200) - Stemirna(SW-BIC-213) Group 2: (N≈200) - Pfizer(BNT162b2) Group 3: (N≈200) -Sinopharm (BIBP) Study groups: There will be three study groups. Study Group Assignment: Randomization (1:1:1) will be applied for subjects to account for the different number of doses per vial for different vaccines and short shelf life.
  Arms: A single 25 μg dose mRNA vaccine SW-BIC-213
Biological: Sinopharm (BIBP);SARS-Cov-2. — The study will be performed in people receiving two doses of Sinopharm vaccine over 180 days (± 30 days) after the second dose prior to enrollment. The three study groups who will receive the booster dose will be assigned as follows:
  Subjects (N≈600) Group 1: (N≈200) - Stemirna(SW-BIC-213) Group 2: (N≈200) - Pfizer(BNT162b2) Group 3: (N≈200) -Sinopharm (BIBP) Study groups: There will be three study groups. Study Group Assignment: Randomization (1:1:1) will be applied for subjects to account for the different number of doses per vial for different vaccines and short shelf life.
  Arms: A third dose of COVID-19 Inactivated vaccine
Biological: Pfizer(BNT162b2);SARS-Cov-2. — The study will be performed in people receiving two doses of Sinopharm vaccine over 180 days (± 30 days) after the second dose prior to enrollment. The three study groups who will receive the booster dose will be assigned as follows:
  Subjects (N≈600) Group 1: (N≈200) - Stemirna(SW-BIC-213) Group 2: (N≈200) - Pfizer(BNT162b2) Group 3: (N≈200) -Sinopharm (BIBP) Study groups: There will be three study groups. Study Group Assignment: Randomization (1:1:1) will be applied for subjects to account for the different number of doses per vial for different vaccines and short shelf life.
  Arms: A single 30μg dose mRNA vaccine Pfizer(BNT162b2)

SUMMARY:
Primary#Objectives #Immunogenicity:To demonstrate the non-inferiority of binding antibody response in terms of geometric mean titers (GMT) of mRNA vaccine compare with mRNA COVID-19 vaccine(Pfizer) 14 days post dose.

Secondary#Immunogenicity:

1. To describe binding antibody profile at D01, D29 and D181 of each study group.
2. To describe the neutralizing antibody profile at D15, D29 and D181 of each study intervention group.

Secondary#Safety:

To assess the reactogenicity and safety of a booster dose in a heterologous vaccination regimen in subjects previously immunized with two Sinopharm doses.

Exploratory#Cell-mediated immunity:

To describe the cellular immune response profile at D01, D08, D15, in a subset of 30 participants for each study group.

Exploratory#Efficacy:

To describe theoccurrence ofvirologically-confirmedCOVID-19 like illness and serologicallyconfirmed SARS-CoV-2 infection.

DETAILED DESCRIPTION:
Endpoint:

Immunogenicity Endpoints:

GMT of Anti-Spike IgG antibody titers will be measured with the ELISA assay on D01, D15.

Immunogenicity Endpoints:

Binding antibody titers to full length SARS-CoV-2 Spike (S) protein will be measured for each study intervention group with the ELISA method.

1. Antibody titer on D01, D29, D181.
2. Fold-rise in antibody titer at D15, D29 and D181 relative to D01Neutralizing antibody titers will be measured with the neutralization assay.
3. Antibody titer on D15, D29 and D181.
4. Fold rise in serum neutralization titer [post/pre] relative to D01 at D15, D29 and D181.

Safety Endpoints:

1. Occurrence of local and systemic AEs reported within 7 days after study vaccination (per group);
2. Occurrence of unsolicited AEs reported within 28 days after study vaccination (per group);
3. Occurrence of SAEs and AESIs within 28 days after study vaccination (per group).

Exploratory#Cell-mediated immunity Endpoints:

INF-γ will be measured in whole blood and/or cryopreserved PBMC following stimulation with pools of S-antigen peptides.

Exploratory#Efficacy Endpoints Occurrence of confirmed symptomatic cases during the study period

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give written informed consent for participation in the study.
2. Male or Female, aged 18 years or above and in good health as determined by study clinician.
3. Female participants of childbearing potential must be willing to ensure that they or their partner use effective contraception from 1 month prior to first immunization continuously until 3months after boost immunization.
4. In the Investigator's opinion, is able and willing to comply with all trial requirements.
5. Subjects had completed the 2-dose series vaccination of COVID-19 inactivated vaccine(Sinopharm) at least 24 weeks with the completed the 2-dose Series as the primary vaccination according to the product label.

Exclusion Criteria:

-

The participant may not enter the study if ANY of the following apply:

1. Confirmed cases, suspected cases or asymptomatic cases of COVID-19;
2. Self-reported history of SARS and MERS infection;
3. Receipt of live attenuated vaccine within one month prior to vaccination and other vaccines within 14 days prior to vaccination;
4. Receipt of any SARS-COV-2 vaccine after last dose of primary vaccination
5. Participants who are pregnant at enrolment or planning to become pregnant during the first 3 months following vaccination
6. Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccines
7. History of allergic disease or reactions likely to be exacerbated by any component of study vaccines
8. Any history of anaphylaxis to any component of vaccine.
9. Bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or continuous use of anticoagulants (warfarin, apixaban, rivaroxaban, dabigatran, edoxaban), or prior history of significant bleeding or bruising following IM injections or venipuncture
10. Suspected or known current alcohol or drug dependency
11. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
12. Severe and/or uncontrolled cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, and neurological illness (mild/moderate well controlled comorbidities are allowed)
13. Scheduled elective surgery during the trial
14. Other reasons investigators did not consider it appropriate to refer to clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2023-06-27 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity | day1, day15
  GMT of Anti-Spike IgG antibody titers will be measured with the ELISA assay on day1 , day 15

CONTACTS AND LOCATIONS:
Overall Officials: Mayfong Mayxay, doctor, Principal Investigator — National Ethics Committee for Health Research(NECHR)
Locations (1):
- Savannakhét Provincial hospital, Savannakhet, Sava, Laos

IPD SHARING:
Plan to Share IPD: No